CLINICAL TRIAL: NCT03536988
Title: Transanal Versus Transabdominal Minimally Invasive Proctectomy With Ileal Pouch-annal Anastomosis On Postoperative Outcomes in Ulcerative Colitis: a Randomized Controlled Trial
Brief Title: TAMIS-IPAA vs. Lap-IPAA for Ulcerative Colitiis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, associate professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JinlingH TAMIS
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-01

CONDITIONS: Ulcerative Colitis; Postoperative Complications; Ileal Pouch
Keywords: Ulcerative Colitiis; Ileal pouch anal anastomosis; Transanal Minimally Invasive Surgery; Postoperative Outcome
MeSH Terms: conditions — Colitis, Ulcerative; Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAMIS-IPAA (Experimental): In TAMIS-IPAA group, transanal minimally invasive surgery of proctectomy with IPAA will be performed.
  Interventions: Procedure: TAMIS-IPAA
- Lap-IPAA (Active Comparator): In Lap-IPAA group, transabdominal minimally invasive surgery of proctectomy with IPAA will be performed.
  Interventions: Procedure: Lap-IPAA

INTERVENTIONS:
Procedure: TAMIS-IPAA — In TAMIS-IPAA group, transanal minimally invasive surgery of IPAA will be performed.
  Arms: TAMIS-IPAA
Procedure: Lap-IPAA — In Lap-IPAA group, transabdominal minimally invasive surgery of IPAA will be performed.
  Arms: Lap-IPAA

SUMMARY:
The objective of this RCT is to compare the postoperative outcome of transanal versus transabdominal minimally invasive proctectomy with ileal pouch-annal anastomosis in patients with ulcerative colitis.

DETAILED DESCRIPTION:
Theoritically, the advantge of TAMIS surgery over traditional trans-abdominal IPAA surgery incudes shorter operation time due to simulatous surgery transanlly and transabdominally, reduced operative difficulty in narrow male pelvis, less retained rectal cuff and less "dog-ear" formation. However, its adgange has not been proven in prospecitve randomized trials. The aim of current study is to compare the short and long-term postoperative outcome of transanal versus transabdominal minimally invasive proctectomy with ileal pouch-annal anastomosis in patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Clincially and pathologically proven ulcerative colitis
* Aged 18-75 years
* Patients who will undergo proctectomy and IPAA surgery, incuding the first stage of two-stage surgery, or the second stage of three-stage or modified two-stage surgery
* Elective surgery
* Informed constent obtained.

Exclusion Criteria:

* A contraindication for minimally invasive surgery or TAMIS surgery
* Ileus or peritonitis
* Previous surgery in rectum
* Pregnancy
* Carcinogenesis of rectum, dysplasia or stricture of ATZ, or planned mucosectomy
* Patients with planned permnant ileostomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications | Day 30
  Postoperative complcations were documented using comprehensive complication index(CCI)

SECONDARY OUTCOMES:
Duration of operation | 24 Hr
  The duration of operation will be documented in minutes, from skin incision to dress coverage
The incidence of pouch extension | 24 Hr
  the need to extend the length of pouch during operation
Intraoperative complications | 24 Hr
  Including anastomotic burst, iatrogenic injury
Estimated blood loss | 24 Hr
  in mLs during surgery
Postoperative anastmotic leakage | Day 90
  Anastomotic leakage was defined as any defect at the anastomotic site confirmed by imaging or during surgical re-intervention, and was categorised according to the impact on clinical management [A, B, C]. Grade A leaks had minimal to no clinical impact on the patient's postoperative course, requiring antibiotics at the most. Grade B leaks required active intervention such as radiological placement of a pelvic drain or transanal lavage. Grade C leaks required re-operation, mostly because the patient was not defunctioned.
Time to GI-2 recovery | Day 90
  Time to GI-2 recovery, a composite end point of the later of upper (first toleration of solid food) and lower (first bowel movement) GI function.
Postoperative length of hospital stay | Day 90
  in days
Overall cost of treatment | up to 1 year
  In Chinese Yuan (CNY)
Remaining length of anal mucosa. | 24 Hr
  The mean lenght of four quadrant during pouchoscopy 2 months after opertion, the length was calculated from the dental line to the anastomotic site.
The incidence of cuffitis and pouchitis | up to 1 year
  Pouchitis is defined as inflammatory condition of the ileal pouch reservoir, while cuffitis is defined as the inflammatory condition of the remnant rectal cuff.
Postoperative quality of life | up to 1 year
  Postoperative quality of life(QoL) is determined using Inflammatory Bowel Disease-Questionaire(IBD-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Gong, Principal Investigator — Jinling Hospital, China
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China